CLINICAL TRIAL: NCT04976166
Title: Shared Decision Making for Choosing renAl Replacement Therapy in Chronic Kidney Disease Patients (SDM-ART Trial)
Brief Title: Shared Decision Making for Choosing renAl Replacement Therapy in Chronic Kidney Disease Patients
Acronym: SDM-ART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sejoong Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDMART
Record Dates: First submitted 2021-06-21; First posted 2021-07-26 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Chronic Kidney Disease Stage 5
Keywords: chronic kidney disease; dialysis; shared decision making
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional group (Active Comparator): Videos and leaflets will be provided. Patients will have education using leaflets for 5 minutes in each hospital at months 0 and 2, respectively.
  Interventions: Behavioral: Education
- Extensive Informed Decision Making group (Experimental): Videos, leaflets, and intensive learning materials will be provided. Patients in the EIDM group will receive more informed and detailed education than those in the conventional group. Patients will have education for more than 10 minutes at months 0 and 2, respectively.
  Interventions: Behavioral: Education
- Shared Decision Making group (Experimental): Videos, leaflets, and intensive learning materials will be provided. Patients will check self-assessment items, and then have education according to the patients' preference using a self-developed counseling calendar. Patients will have education for more than 10 minutes at months 0 and 2, respectively.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — More informed and detailed education
  Arms: Extensive Informed Decision Making group
Behavioral: Education — Shared decision making
  Arms: Shared Decision Making group
Behavioral: Education — education as usual
  Arms: Conventional group

SUMMARY:
Shared decision making (SDM) is an approach where clinicians and patients make decisions together using the best available evidence. An understanding of the patient's treatment goals, the advantages and disadvantages of treatment options, and the likelihood of achieving the outcomes are important to patients. International guidelines recommend that all patients with chronic kidney disease (CKD) at pre-dialysis stage should be educated to improve their knowledge and understanding of their condition and to choose the options for renal replacement therapy (RRT).

Despite these recommendations, pre-dialysis educations are often infrequent. Many patients feel unprepared. Wrong or insufficient understanding due to insufficient explanation of treatment can lead to negative emotions. This may lead to a situation in which the patient loses the opportunity to make patient's own choices, resulting in emergency dialysis or dialysis modality that is not suitable for patients. Therefore, this study aims to evaluate whether SDM has an effect on the choice of RRT among CKD patients.

DETAILED DESCRIPTION:
This study will be conducted as a multicenter, open-label, randomized, pragmatic clinical trial. A total of 1,194 participants with CKD considering RRT will be randomized into 3 groups. Patients in the conventional group will have education using leaflets. Patients in the extensive informed decision making (EIDM) group will receive more detailed education using intensive learning materials than those in the conventional group. Shared decision making (SDM) group patients will have education according to questionnaires of self-assessment items using a self-developed counseling calendar.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease whose nephrologist predicts initiation of renal replacement therapy within 12 months:

  1. Patients with grade 5 of chronic kidney disease [defined as a creatinine-based estimated glomerular filtration rate (eGFR) < 15 ml/dL/1.73m2 at least 2 times at intervals of 2 weeks or longer]
  2. Patients with the cystatin C-based eGFR < 15 ml/dL/1.73m2 at least once if the creatinine-based eGFR does not accurately evaluate the kidney function of patient due to patient characteristics
  3. Patients whose nephrologist require renal replacement therapy within 12 months due to the patient's comorbidities even when the eGFR is 15ml/dL/1.73m2 or higher
* Patients aged between 19 and 80 years
* Patients who understand the study
* Patients who have no permanent access device for long-term maintenance dialysis

Exclusion Criteria:

* Patients who have contraindication to perform peritoneal dialysis due to abdominal surgery
* Patients whose life expectancy is less than 6 months due to underlying diseases
* Patients who have enrolled in other clinical trials within 3 months or plan to participate in other clinical trials during this clinical trial period
* Patients judged by the investigator to be inappropriate for participation in this clinical trial

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1194 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The ratio of hemodialysis to non-hemodialysis | 12 months
  To compare the proportion of hemodialysis versus non-hemodialysis (peritoneal dialysis and kidney transplantation) treatments among the groups

SECONDARY OUTCOMES:
Economic efficiency using a cost-utility analysis | Month 2, and 12
  The incremental cost-utility ratio (ICUR) is calculated by the ratio of differences in costs and utilities.
Patients' satisfaction assessed by Patient Satisfaction Questionnaire (ZUF-8) | Month 0, 2, and 12
  The ZUF-8 is an 8-items questionnaire to assess satisfaction in patients using a scale from 1,"poor" to 4,"excellent". Originally, ZUF-8 used a 4-point scale, but in this study, the investigators further extended the scoring system of this questionnaire from four to five incremental stages of perceived satisfaction, i.e. "poor (1)," rather good (2)," good (3)," very good (4)," extraordinary (5)". The minimum value is 8 and the maximum value is 40. Higher scores mean a better outcome.
Patients' evaluation of the SDM process assessed by Shared Decision-Making Questionnaire (SDM-Q-9) | Month 0, 2, and 12
  The SDM-Q-9 questionnaire is a nine item measure. Items are reported with six response options ranging from 0, "completely disagree", to 5, "completely agree". In this study, six response options were converted into five incremental stages, i.e. "strongly disagree (1)," somewhat disagree (2)," neither disagree nor agree (3)," somewhat agree (4)," strongly agree (5)". To calculate the total scale score, items are summed resulting in a range from 9-45. Higher scores reflect a participant's participation in shared decision making regarding their treatment.
Patients' adherence to medication assessed by Morisky 8-item Medication Adherence Scale (MMAS-8) | Month 0, 2, and 12
  The MMAS-8 is an 8-items questionnaire and the scale included 7 items with yes/no response options and 1 item with a 5-point Likert scale response option. Cumulative score based on 8 items are used to obtain final adherence score ranging from 0 to 8. Adherence is defined accordingly as low (score 0-5), medium (score 6-7) and high (score 8).
unplanned dialysis | 12 months
  To compare the rate of unplanned dialysis among the groups

CONTACTS AND LOCATIONS:
Overall Officials: Sejoong Sejoong, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (19):
- South Korea (19):
  - Bundang Seoul National University Hospital, Seongnam-si, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Daejeon Eulji Medical Center, Daejeon
  - Dongguk University Ilsan Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Pusan National University Hospital, Pusan
  - Ewha Woman's University Seoul Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea Eunpyeong St. Mary's Hospital, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: No